CLINICAL TRIAL: NCT04746456
Title: Vulvovaginal Atrophy Questionnaire (VVAQ): Psychometric Validation of a Novel Patient Reported Outcome Measure (PROM)
Brief Title: Vulvovaginal Atrophy Questionnaire (VVAQ): Psychometric Validation of a Novel PROM
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jan Shifren, MD, Director, Midlife Women's Health Center, Dept. Ob/Gyn, Massachusetts General Hospital
Other Study IDs: 2020P003777
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Vulvovaginal Atrophy; Menopause; Genitourinary Syndrome of Menopause
Keywords: Vulvovaginal atrophy; Menopause; Genitourinary Syndrome of Menopause; Patient Reported Outcome Measure (PROM)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Menopausal women: Women will complete a series of questionnaires, including the VVAQ

SUMMARY:
The goal of this study is to perform a quantitative assessment of the psychometric properties of the Vulvovaginal Atrophy Questionnaire (VVAQ), a novel patient reported outcome measure (PROM), through a REDCap survey of menopausal women with and without symptomatic vulvovaginal atrophy (VVA)/genitourinary syndrome of menopause (GSM).

DETAILED DESCRIPTION:
Bothersome vaginal dryness, dyspareunia, urinary symptoms, and related sexual and quality of life sequelae are common problems for women during and after the menopausal transition. These genitourinary symptoms adversely affect the lives of menopausal women, impacting daily activities, emotional wellbeing, sexual function, and interpersonal relationships. Genitourinary syndrome of menopause (GSM) describes anatomical changes and bothersome symptoms associated with menopausal estrogen deficiency involving the labia, vagina, urethra, and bladder. Symptoms must be bothersome and not accounted for by another diagnosis. Vulvovaginal atrophy (VVA) is a component of GSM. Despite effective and safe therapeutic options for symptomatic VVA/GSM, many women remain untreated. Although vulvovaginal symptoms are commonly reported in community-based studies of menopausal women, the lack of a validated measure of symptomatic VVA/GSM has limited our ability to accurately quantify its prevalence, predictive factors, and associated outcomes. Using ad hoc or non-validated survey questions, past studies have reported vulvovaginal symptoms in 27-85% of menopausal women. Despite the broad sampling and diverse populations included in these studies, the absence of a validated measurement tool limits our understanding of the true prevalence and predictors of this disorder.

A new patient reported outcome measure (PROM), the Vulvovaginal Atrophy Questionnaire (VVAQ), is under development in a collaboration between the Massachusetts General Hospital Midlife Women's Health Center and the North American Menopause Society (NAMS) to provide a validated measure for assessing symptomatic VVA/GSM. Significant advances in research and improved patient care are anticipated from availability of a brief, validated PROM for evaluating symptomatic VVA/GSM in menopausal women. Self-administered questionnaires and brief symptom scales for other common problems affecting women, including vasomotor symptoms, insomnia, overactive bladder, and sexual dysfunction have greatly impacted the way research studies are performed and clinical problems addressed in midlife women. The VVAQ is being developed for use both in clinical and epidemiological research and patient care settings, with the goal of advancing knowledge about symptomatic VVA/GSM and improving the care of menopausal women. A validated measure for assessing symptomatic VVA/GSM and response to treatment interventions, freely available in the public domain, will provide a critical research tool for epidemiologic studies and efficacy assessment in clinical trials of new therapies. A validated PROM will provide clinicians from multiple specialties and researchers from a wide range of fields with a practical and efficient means for assessing symptomatic VVA/GSM in midlife women.

This is an observational psychometric validation study through a REDCap survey of approximately 200 menopausal women age 45 years or older with and without symptomatic VVA/GSM. No medications or treatments will be administered. Appropriate Human Research Committee review and approval was obtained prior to study initiation. Potential study participants will be identified during regularly scheduled office visits for routine clinical care by a select group of approximately 20 clinicians with expertise in the care of menopausal women. These clinicians all will be members of the North American Menopause Society (NAMS) who have agreed to serve as NAMS VVAQ Referring Clinicians. Appropriateness for referral to the study will be confirmed by the NAMS VVAQ Referring Clinician at the time of routine patient care visits. At the end of a clinic visit, a NAMS VVAQ Referring Clinician will determine if a patient is eligible to be referred to the study.

Potential Participants informed about the study by a NAMS VVAQ Referring Clinician will then log in to the study's secure REDCap website and review information about the study. If interested, participants will consent to study participation and complete the study questionnaires. Participants will be informed that researchers associated with the North American Menopause Society (NAMS) and the Massachusetts General Hospital (MGH) Midlife Women's Health Center are studying the genitourinary syndrome of menopause (GSM), a condition that affects women after menopause and includes vaginal dryness and pain with sexual activity. To learn more about GSM, researchers will be studying menopausal women both with and without this problem. Women are eligible to participate if they are menopausal, age 45 years or older, and have been referred to the study by their health care provider after an office visit that included a pelvic exam. Participation involves completing questionnaires at home through a secure website on a computer within 2 weeks of their office visit. Completing the questionnaires will take approximately 25 minutes.

Participants will be informed that they will be identified only by a study identification number on the questionnaires. No identifying information will be collected, including name or date of birth. As researchers will need to know whether a participant's clinician saw evidence of vulvovaginal atrophy on a recent pelvic exam, participants will enter into the secure study website information provided to the participant by the NAMS VVAQ Referring Clinician regarding pelvic exam findings, including degree of vulvovaginal atrophy and evidence of a urogenital condition unrelated to menopausal estrogen deficiency. Participants who complete the survey will be given the option of completing the questionnaires a second time 2 weeks later. This option will end after 50 participants have completed the "re-test' part of the study.

The statistical analyses and tests outlined below will be used to assess the psychometric properties of the VVAQ. If the VVAQ is found to be multi-dimensional (i.e., having multiple factors or independent domains), analyses will be performed separately on each factor or domain, in addition to comparisons for the overall scale. A quantitative scoring algorithm will be developed and tested for sensitivity and specificity. Comparisons across groups (women with and without symptomatic VVA) will be performed to establish discriminant validity. Inter-item and test-retest reliability will be ascertained from responses in participants with and without symptomatic VVA. Factor analysis will be performed in the group of women with symptomatic VVA and for all participants combined (to ensure adequate sample size), and discriminant validity testing will be done across all items and factor scores. Convergent validity will be assessed by examining correlations between item and factor scores, as well as factor and item scores. Statistical Analyses: 1) Item Analysis, 2) Item Reduction, 3) Scoring Algorithm, 4) Exploratory Factor Analysis, 5) Item Response Theory Analysis, 6) Internal Consistency, 7) Factor Structure & Final Scoring Algorithm, 8) Test-Retest Reliability, 9) Convergent/Divergent Validity, 10) Discriminant (Known Groups) Validity.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age > 45 years
* Menopausal, defined as: > 1 year since last menses (with a uterus, without progestin- releasing IUD, without prior endometrial ablation), or > 6 months since bilateral oophorectomy
* Pelvic exam completed as part of visit
* Able to communicate in English

Exclusion Criteria:

* Chronic, bothersome vaginal symptoms before menopause (e.g. vulvar or vaginal pain, dryness, itching, discharge, discomfort with sexual activity)
* History of chronic urogenital condition (vulvar, vaginal, urinary), involving pain, pruritis, discharge, or inflammation, unrelated to menopausal estrogen deficiency
* History of lichen sclerosis or lichen planus
* History of vulvar, vaginal or cervical cancer
* Prior vulvar or vaginal surgery (office biopsy allowed)
* Active major medical illness (e.g., unstable heart disease, untreated psychiatric disorder) that might interfere with the ability to participate in the study
* Undiagnosed vaginal bleeding
* Exam findings consistent with a urogenital condition unrelated to menopausal estrogen deficiency (e.g. yeast or BV vaginitis, vulvodynia, vulvo-vestibulitis, lichen sclerosis, lichen planus)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: This is an observational psychometric validation study through a REDCap survey of approximately 200 menopausal women age 45 years or older with and without symptomatic VVA/GSM. No medications or treatments will be administered.
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Responses to VVAQ and additional relevant questionnaires | Baseline
  Results of REDCap survey

CONTACTS AND LOCATIONS:
Overall Officials: Jan Shifren, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Shifren JL, Zincavage R, Cho EL, Magnavita A, Portman DJ, Krychman ML, Simon JA, Kingsberg SA, Rosen RC. Women's experience of vulvovaginal symptoms associated with menopause. Menopause. 2019 Apr;26(4):341-349. doi: 10.1097/GME.0000000000001275. PMID 30531443